CLINICAL TRIAL: NCT02139657
Title: An Open-label, Single-arm Study to Evaluate the Safety and Antibody Titers Specific to the Rabies Virus in Healthy Subjects After Receiving a Single Dose of Intramuscularly Administered Rabies Immune Globulin (Human)
Brief Title: An Open-label, Single-Arm Study to Evaluate the Safety and Rabies Virus Antibody Titers of Intramuscularly Administered Rabies Immune Globulin (Human)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Grifols Therapeutics LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GTI1301
Record Dates: First submitted 2014-04-28; First posted 2014-05-15 (Estimated); Last update posted 2014-07-24 (Estimated); Status verified 2014-07

CONDITIONS: Rabies
Keywords: Rabies; Rabies virus; Rhabdoviridae; Rabies immune globulin; Rabies antibodies; Passive rabies immunization
MeSH Terms: conditions — Rabies | interventions — Caprylates

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- RIG-C (Experimental): Single 20 IU/kg dose of RIG-C by intramuscular injection
  Interventions: Biological: RIG-C

INTERVENTIONS:
Biological: RIG-C
  Other Names: Rabies Immune Globulin (Human), Caprylate/Chromatography Purified

SUMMARY:
This is a single-arm, open-label study of Rabies Immune Globulin (Human), Caprylate/Chromatography Purified (RIG-C), in approximately 12 healthy subjects. The purpose of this study is to characterize the rabies virus-specific antibody titer after a single intramuscular injection of 20 IU/kg RIG-C and to evaluate the safety and tolerability of RIG-C.

ELIGIBILITY:
Inclusion Criteria:

* In good health in the judgment of the Investigator as determined by medical history, physical examination, and screening laboratory assessments.
* Female of childbearing potential must have a negative result on the screening serum pregnancy test and must agree to practice contraception by a method of proven reliability (includes abstinence) for the duration of the study.

Exclusion Criteria:

* Pregnant or lactating females.
* Clinical evidence of any significant acute or chronic disease that may interfere with successful completion of the trial.
* Clinically significant history of the following: cardiovascular disease, hyperlipidemia, serious respiratory disease including bronchitis or asthma, endocrine disorder, liver disease, glaucoma, gastrointestinal disease, disorder of the reticuloendothelial system, or neurologic illness.
* History of angioedema or nephrotic syndrome.
* Non-controlled arterial hypertension.
* Anemia at screening.
* Significant proteinuria (> 1 + on urine dipstick) and/or has a history of acute renal failure and/or severe renal impairment or a blood urea nitrogen or creatinine more than 2.5 times the upper limit of normal at screening and/or currently receiving dialysis.
* Elevated liver enzymes (aspartate transaminase, alanine aminotransferase) and Gamma-glutamyl Transferase) equal to or greater than 1.5 times the upper limit at screening.
* Previously received the rabies vaccine and/or rabies immune globulin.
* Received infusion of a blood/plasma product or fraction within the past 12 months, including any type of immune globulin.
* Known adverse reaction to administration of any immune globulin or other blood/plasma products.
* Experienced anaphylactic shock with the administration of blood/plasma products.
* Known medical history of selective immunoglobulin A (IgA) deficiency.
* Received any corticosteroids, immunosuppressants, or immunomodulators within 6 weeks prior to screening.
* Expects to receive oral or topical non-steroidal anti-inflammatory drugs (NSAIDs), acetaminophen, antihypertensives, and/or antihistamines 24 hours before or after investigational product administration during the Baseline/Treatment, Study Day 0 visit.
* Currently receiving any anti-viral treatment.
* Screening laboratory results indicative of an acute or chronic infection with hepatitis A virus (HAV), hepatitis B virus (HBV), hepatitis C virus (HCV), human immunodeficiency virus (HIV), or parvovirus B19 (B19V).
* Participated in another clinical trial within 30 days prior to screening (imaging studies without investigative treatments are permitted) or has received any investigational products within the previous 3 months.
* Not willing to postpone receiving any live virus vaccines until 3 months after receiving investigational product.
* History of a psychiatric illness requiring hospitalization.
* Known substance or prescription drug abuse in the past 12 months.
* Any active medical illness that the Investigator may consider a potential confounding condition that would interfere with the study visits and/or procedures.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2014-03; Primary Completion 2014-05 (Actual); Study Completion 2014-05 (Actual)

PRIMARY OUTCOMES:
Rabies Virus Antibody Titer | 10 days post-RIG-C dosing

SECONDARY OUTCOMES:
Number of subjects who discontinue due to adverse events | 21 days

CONTACTS AND LOCATIONS:
Locations (1):
- Tempe, Arizona, United States

REFERENCES:
- [Derived] Hanna K, Cruz MC, Mondou E, Corsi E, Vandeberg P. Safety and neutralizing rabies antibody in healthy subjects given a single dose of rabies immune globulin caprylate/chromatography purified. Clin Pharmacol. 2018 Jun 26;10:79-88. doi: 10.2147/CPAA.S166454. eCollection 2018. PMID 29983597